CLINICAL TRIAL: NCT01744002
Title: The Addition of Cervical Unilateral Posterior Anterior Mobilization (UPA) in the Treatment of Patients With Shoulder Impingement Syndrome: A Randomized Clinical Trial
Brief Title: Neck Mobs and Impingement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Walsh University (Other)
Responsible Party: Principal Investigator, Chad Cook, Principal Investigator, Walsh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12812
Record Dates: First submitted 2012-12-02; First posted 2012-12-06 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2012-12

CONDITIONS: Shoulder and Neck
Keywords: Shoulder, Impingement syndrome, Neck

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shoulder Treatment with Neck Mobilization (Experimental): The experiment group will receive shoulder treatment with an emphasis on 1) range of motion activities, 2) joint mobilization, 3) rotator cuff strengthening and 4) a home exercise program that consists of shoulder strengthening exercises; and Unlateral Posterior Anterior Mobilization to the cervical spine; applied as 3 X 30 seconds, to each comparable (stiff or painful) segment.
  Interventions: Other: Shoulder treatment and neck mobilization
- Control Group (Active Comparator): The control group will receive shoulder treatment with an emphasis on 1) range of motion activities, 2) joint mobilization, 3) rotator cuff strengthening and 4) a home exercise program that consists of shoulder strengthening exercises.
  Interventions: Other: Control

INTERVENTIONS:
Other: Shoulder treatment and neck mobilization — This group will receive shoulder treatment with an emphasis on 1) range of motion activities, 2) joint mobilization, 3) rotator cuff strengthening and 4) a home exercise program that consists of shoulder strengthening exercises; and joint mobilizations to the neck.
  Arms: Shoulder Treatment with Neck Mobilization
Other: Control — This group will receive shoulder treatment with an emphasis on 1) range of motion activities, 2) joint mobilization, 3) rotator cuff strengthening and 4) a home exercise program that consists of shoulder strengthening exercises.
  Arms: Control Group

SUMMARY:
The objective of this study is to investigate whether treatment directed at the neck and shoulder is more beneficial than treatment directed solely at the shoulder; for patients with shoulder impingement syndrome.

(The hypothesis is that patients who receive neck mobilization will improve at a more significant rate than those who do not receive neck mobilization)

DETAILED DESCRIPTION:
All treatment will be provided by licensed physical therapist within the United States. The clinicians affiliated with this study have experience in data collection and have participated in a recent trial that was sponsored by Walsh University.

At baseline, after consent for the study, patients will be randomized into two groups: 1) shoulder treatment and active mobilization to the neck and 2) shoulder treatment and placebo mobilization to the neck. Baseline data will be collected including all self-report measures.

Both groups will receive shoulder treatment with an emphasis on 1) range of motion activities, 2) joint mobilization, 3) rotator cuff strengthening and 4) a home exercise program that consists of shoulder strengthening exercises. The active neck group will receive UPA's to the cervical spine; applied as 3 X 30 seconds, to each comparable (stiff or painful) segment. The physical therapist will place their hands on the neck of the patient for the placebo group but will not perform the oscillations that are characteristic of mobilization.

All patients will receive a home program designed to increase range of motion and strength. None of the home program focused exercises will be targeted to the neck. The shoulder exercises will be tailored to each specific patient and will not be standardized.

Patients will be treated for the duration of their care using the same foci (1) range of motion activities, 2) joint mobilization, 3) rotator cuff strengthening and 4) a home exercise program that consists of shoulder strengthening exercises). The length of the treatment will be determined by the progress of the patient and by the attending therapist.

ELIGIBILITY:
Inclusion Criteria:

* Patients, age 18 and older, with shoulder impingement syndrome, who attend care at a physical therapy outpatient setting, will be screened for eligibility for the study by the treating physical therapists. For patients to meet inclusion requirements, they require the following:

  1. Report pain or dysfunction with elevated (overhead) arm activities, Demonstrate pain during active shoulder movements
  2. Demonstrate a positive Neer or Hawkins Kennedy Test
  3. Report an onset that is non-traumatic
  4. Report an onset within the last 12 months
  5. Demonstrate a painful arc of movement during forward elevation of the arm from 60° to 120°

Exclusion Criteria:

* Exclusion criteria will include The presence of any red flags (i.e., tumor, metabolic diseases, rheumatoid arthritis, osteoporosis, prolonged history of steroid use, etc.), a history of frozen shoulder, disorders of the acromioclavicular joint, degenerative arthritis of the glenohumeral joint, calcifying tendonitis, shoulder instability, posttraumatic disorders, or shoulder surgery and/or elbow, hand, wrist and blatantly misdiagnosed cervical spine disorders (e.g., cervical radiculopathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Quick Disabilities of Shoulder and Hand Questionaire (QuickDASH) | participants will be followed for the duration of the treatment which is on average 4 weeks
  The QuickDASH is a shortened version of the DASH Outcome Measure. Instead of 30 items, the QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. The tool has been validated and has similar psychometric properties to the DASH

SECONDARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | participants will be followed for the duration of the treatment which is on average 4 weeks
  The NPRS will be used to capture the patient's level of pain. Patients will be asked to indicate the intensity of current, best, and worst levels of pain over the past 24 hours, using an 11-point scale ranging from 0 "no pain" to 10 "worst pain imaginable." The average of the 3 ratings will be used to represent the patient's level of pain over the previous 24 hours.

OTHER OUTCOMES:
Patient Acceptable Symptom State (PASS) | participants will be followed for the duration of the treatment which is on average 4 weeks
  The PASS is the symptom state in which the patients feel that their current well-being is acceptable. The question is dichotomous (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Cook, PhD, Principal Investigator — Walsh U
Locations (1):
- Walsh University, North Canton, Ohio, United States